CLINICAL TRIAL: NCT00120497
Title: Growth Hormone and Insulin Resistance in Children With Intrauterine Growth Restriction
Brief Title: Study to Examine Insulin Resistance During Growth Hormone Treatment for Short Stature Due to Low Birthweight
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Lynne L. Levitsky, M.D., Massachusetts General Hospital
Other Study IDs: 2005P-000384; IRG 2004-0964
Record Dates: First submitted 2005-07-13; First posted 2005-07-18 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Fetal Growth Retardation
Keywords: short stature; intrauterine growth restriction; insulin resistance; intramyocellular lipid; small for gestational age; glucose tolerance
MeSH Terms: conditions — Fetal Growth Retardation; Dwarfism; Insulin Resistance | interventions — Human Growth Hormone; DNA, Ribosomal; Growth Hormone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: somatropin (rDNA) — Dosage form/strength: 13.8 mg powder in 2-chamber cartridge; reconstitutes to 10 mg/ml
  Dosage regimen: 0.48 mg/kg/week
  Route/rate of administration: subcutaneous injection, daily dose
  Other Names: Genotropin; recombinant human growth hormone

SUMMARY:
Insulin resistance is common among children with low birthweight. Moreover, growth hormone treatment for ensuing short stature also causes insulin resistance. Our objective is to examine these processes. Insulin resistance has recently been linked to the accumulation of stores of fat in muscle cells which can be measured by MRI. We hypothesize that children who are short due to low birthweight have increased muscle fat stores, but that growth hormone treatment will paradoxically reverse this association. To test this hypothesis, muscle fat stores will be measured in children who are short due to low birthweight before and after receiving growth hormone therapy. Other parameters linked to insulin resistance (glucose tolerance, blood markers, and body composition) will also be assessed. This study may lead to ways to increase growth hormone safety and dose limitations.

DETAILED DESCRIPTION:
Growth hormone (GH) is an effective height-enhancing treatment for short stature. One underlying disorder is intrauterine growth restriction (IUGR). Increased growth enhances quality of life as well as improving body composition, metabolism, and lipid distribution. However, both GH therapy and IUGR can cause insulin resistance. Scientists have recently linked insulin resistance to the accumulation of fat inside muscle cells (intramyocellular lipids or IMCL). Although GH generally reduces overall body fat, its effect on IMCL has not yet been examined. This association can be examined in children with IUGR initiating GH treatment for short stature.

Hypothesis: Children with IUGR will have increased IMCL linked to insulin resistance, but GH treatment may paradoxically reverse this association.

Objectives: To assess changes in IMCL during GH therapy and to increase our knowledge of GH action.

Study design: Prepubertal children initiating a course of GH therapy indicated by persistent short stature as a result of IUGR will be recruited to participate in a crossover study.

* IMCL (soleus and tibialis anterior) will be measured non-invasively by proton magnetic resonance spectroscopy (1H-MRS)
* Body composition will be measured by DEXA and morphometry
* Whole body insulin sensitivity (IS) will be assessed by oral glucose tolerance
* Levels of plasma lipids and hormones will be measured

Endpoints: The primary endpoint will be to define the effect of GH on IMCL content in IUGR children. Secondary endpoints will be (i) to compare the relationships between IMCL and IS before and after GH therapy, and (ii) to identify the correlative changes in plasma hormones and metabolites that may underlie the IMCL changes.

Significance: IMCL is anticipated to be a valuable probe for understanding GH effects on glucose homeostasis. This study is intended to reveal strategies for enhancing GH efficacy without compromising IS. New pharmacological approaches to manage GH-induced glucose intolerance would be important in counteracting this limiting factor in GH dosing.

ELIGIBILITY:
Inclusion Criteria:

* height < 5%-ile
* birthweight < 10%-ile for gestational age
* gestation: ≥ 36 weeks
* male or female
* age: 8-12 years
* BMI = 10-90%-ile
* normal childhood activity, no physical or other limitations
* bone age ≤ 12 years
* normal, balanced diet (20-40% calories from fat)

Exclusion Criteria:

* puberty (beyond Tanner Stage 1)
* diabetes in subject or first degree relative
* sex steroid therapy
* chronic conditions requiring medication
* other causes of short stature (e.g., Prader-Willi, intracranial lesions, hypopituitarism, Turner syndrome, GHD, etc.)
* significant systemic disease (pulmonary, cardiac, renal, or other)
* non-removable metal
* other conditions judged by the investigator to pose a hazard (including history of neoplasm)
* simultaneous participation in another medical investigation or trial

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, age 6-12 years old, with short stature associated with low birth weight
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2005-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne L Levitsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States